CLINICAL TRIAL: NCT02963272
Title: Interest of ST2 to Diagnosis and Management of Patients With Heart Failure (HF)
Brief Title: ST2 for the Management of Heart Failure - STADE-HF
Acronym: STADE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL16_0194; 2016-A01148-43 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-10-31; First posted 2016-11-15 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure; Diastolic Heart Failure; Systolic Heart Failure Stage C
Keywords: Heart failure; ST2; fibrosis
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional strategy (Other): Conventional strategy to manage the patients with HF, following the international guidelines
  Interventions: Other: Conventional strategy
- ST2-guided strategy (Other): Management of patients follow the international guidelines but are also guided by the ST2, to adapt the drugs indicated in patients with HF.
  Interventions: Other: ST2-guided strategy

INTERVENTIONS:
Other: Conventional strategy — Conventional strategy to manage the patients with HF, following the international guidelines.
  Arms: Conventional strategy
Other: ST2-guided strategy — patients wit ST2 over the median are targeted with higher doses of drugs with putative effects on fibrosis and anti HF pathophysiology
  Arms: ST2-guided strategy

SUMMARY:
Heart failure (HF) is a severe disease, burdened with a poor prognosis (30% mortality at 2 years, 30% of rehospitalization within 1 month). It is also a major cause of health burden representing between 1.5 and 2 billions euros per year in France. Approximately 75% of these costs are due to hospitalization.

Besides physical examination and echocardiography, biology may help refine the diagnosis, but also could provide powerful prognostic parameters.

This study aims to assess the value of ST2 in the management of patients admitted for HF to reduce readmission at one month.

DETAILED DESCRIPTION:
Background and rationale:

Heart failure (HF) is a severe disease, burdened with a poor prognosis (30% mortality at 2 years, 30% of rehospitalization within 1 month). It is also a major cause of health burden representing between 1.5 and 2 billions euros per year in France. Approximately 75% of these costs are due to hospitalization.

Besides physical examination and echocardiography, biology may help refine the diagnosis, but also could provide powerful prognostic parameters. The natriuretic peptides are already available and widely used to this purpose. Other biomarkers such as fibrosis markers are promising. In a recently published preliminary work of a cohort of 180 cardiac patients, ST2 is proving to be a powerful prognostic biomarker.

This study aims to assess the value of ST2 in the management of patients admitted for HF to reduce readmission at one month.

Primary and secondary endpoints:

Primary endpoint:

- Interest of ST2 to decrease rehospitalization at one month in patients admitted for HF in the cardiology department and / or Internal Medicine.

Secondary objective:

* economic evaluation
* Clinical Target: mortality, stay at hospital duration
* Impact on biological markers of HF, renal function Population: Any adult being hospitalized for any type of HF. A total of 300 patients will be over a period of 36 months, divided into 2 arms.

Methods: interventional, randomized, opened: the two strategies "ST2 available" versus "ST2 not available" will be compared The duration of patient participation is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure hospitalization

Exclusion Criteria:

* Other study
* Pregnancy, feeding
* Refusal
* Not possible to perform information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Rehospitalization | 1 month
  The frequence of the rehospitalization of the patient according to the treatment received

SECONDARY OUTCOMES:
Economic evaluation | 1 month and 1 year
  Compare the hospitalization cost at 1 month and the cost of biological diagnostic strategies (NT-proBNP with or without ST2)
Mortality | 1 month and 1 year
  measure of mortality
Biological markers of HF Assay | 1 month and 1 year
  Measure of biological marker ST2
Stay at hospital duration | 1 month and 1 year
  Evaluation of duration of hospitalisation
Markers of the renal function assay | 1 month and 1 year
  Measure of biological marker of renal function
Rehospitalization for heart failure | 1 month and 1 year
  Rehospitalization rate for heart failure
Rehospitalization for all causes | 1 month and 1 year
  Rehospitalization rate for all causes

CONTACTS AND LOCATIONS:
Overall Officials: François ROUBILLE, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Regional Hospital Arnaud de Villeneuve, Montpellier, Languedoc-Roussillon, France

IPD SHARING:
Plan to Share IPD: No